CLINICAL TRIAL: NCT03959631
Title: Effectiveness and Cost-effectiveness of a Virtual Intervention (VCoP) to Improve the Empowerment of Patients With Ischaemic Heart Disease in Primary Care: Cluster Randomized Controlled Trial
Brief Title: Effectiveness and Cost-effectiveness of a VCoP to Empowerment of Patients With Ischaemic Heart Disease in PHC: Cluster-RCT
Acronym: Empodera-dos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gerencia de Atención Primaria, Madrid (Other Government)
Collaborators: Avedis Donabedian Research Institute (Other); Servicio Canario de Salud (Other)
Responsible Party: Principal Investigator, Sofia Garrido Elustondo, Epidemiologist, Gerencia de Atención Primaria, Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: PI18/01397; PI18/01333 (Other Grant/Funding Number: Servicio de Evaluación del Servicio canario de la Salud); PI 18/01404 (Other Grant/Funding Number: Avedis Donabedian Research Institute)
Record Dates: First submitted 2019-05-13; First posted 2019-05-22 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Ischemic Heart Disease Chronic
Keywords: Ischemic Heart Disease Virtual Community of Practice empowerment

STUDY DESIGN:
Intervention Model Description: Design: pragmatic randomized controlled trial, with two parallel arms, multicenter, 18 months of follow-up
  Setting Primary Care Centres belonging to the Autonomous Communities of Catalonia, (329), Madrid (262) and the Canary Islands (102).
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigator and outcomes Assessor don´t Know the intervention assigned to each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The intervention group will be offered participation for 6 months in a Virtual Communities of practice based on a web 2.0 platform in which there is interaction with other patients and with a multidisciplinary team of professionals. The intervention will be co-designed with a group of patients and a group of primary and specialized care professionals.
  Interventions: Behavioral: Virtual Communities of practice
- Control group (No Intervention): The control group will not receive any specific intervention. They receive usual care according to actually clinical practice guidelines.

INTERVENTIONS:
Behavioral: Virtual Communities of practice — based on a web 2.0 platform in which there is interaction with other patients and with a multidisciplinary team of professionals. The intervention will be co-designed with a group of patients and a group of primary and specialized care professionals.
  Arms: Intervention group

SUMMARY:
Objective: to evaluate the effectiveness and estimate the costs of a Virtual Community of Practice in the improvement of the activation of patients with Ischemic Heart Disease in Primary Care .

Methods:

Design: pragmatic randomized controlled multicentric trial. Setting: health centres belonging to the Autonomous Communities of Catalonia, Madrid and the Canary Islands. Population: 246 patients with Ischemic Heart Disease in Primary Care. Randomization: randomization will be central and automatically performed by the online "e-mpodera" platform and the assigned group will be communicated to the patient once he or she has entered the platform and completed baseline assessment. Intervention: the intervention group will be offered participation for 6 months in a Virtual Community of Practice based on a web 2.0 platform in which there is interaction with other patients and with a multidisciplinary team of professionals. The intervention will be co-designed with a group of patients and a group of primary and specialized care professionals. The control group will receive usual care. Measurements: the main variable will be measured using the Patient Activation Measure questionnaire at baseline, 6, 12 and 18 months. Secondary variables: sociodemographic and clinical variables of the patients; knowledge test (questionnaire of risk cardiovascular factories , attitudes (Self-efficacy Managing Chronic Disease Scale ), adherence to Mediterranean diet (Mediterranean Diet), level of physical activity (International Physical Activity Questionnaire), medication adherence (Adherence Refill and Medication Scale (ARMS-e), depression (Patient Health Questionnaire), anxiety (Hospital Anxiety and Depression Scale), quality of life (EQ-5D-5L); variables related to the use of health resources; variables related to the use of the Virtual Community of Practice . Data will be collected from self-reported questionnaires and the electronic medical records. Analysis: a linear regression model of mixed effects will be estimated to estimate the effect of participating in the Virtual Community of Practice. In addition, subgroup analyses will be carried out and indicators of the functioning of the Virtual Community of Practice will be measured through techniques of Social Network Analysis and Control Charts. There will be an economic evaluation of the Virtual Community of Practice from the perspective of the National Health System and from the social perspective.

DETAILED DESCRIPTION:
Methods:

Design: pragmatic randomized controlled trial, with two parallel arms, multicenter, 18 months of follow-up.

Time Frame: 18 months.

Setting Primary Care Centres belonging to the Autonomous Communities of Catalonia, (329), Madrid (262) and the Canary Islands (102).

Study Population: patients with a recent diagnosis of ischemic heart disease in follow-up by Primary Care (diagnosis of ischemic heart disease in the year prior to inclusion in the study).

Inclusion criteria: age over 18 years; Active diagnosis of ischemic heart disease in the year prior to inclusion in the study; have Internet at home or phone; be able to follow the requirements of the study; having signed informed consent for participation in the study.

Exclusion criteria: low probability of cooperation in the study, bystanders or displaced status, institutionalized, with a terminal illness, physical or mental disability that prevents respond to questionnaires properly.

Population: 246 patients with Heart Disease in Primary Care. (123 patients per arm) .

Randomization: patients will be randomly assigned to the intervention (VCoP) or control group. The randomization will be central and automatically performed by the online "e-mpodera" platform and the assigned group will be communicated to the patient once he or she has entered the platform and completed baseline assessment.

Intervention:

* The intervention group will be offered participation for 6 months in a Virtual Community of Practice based on a web 2.0 platform in which there is interaction with other patients and with a multidisciplinary team of professionals. The intervention will be co-designed with a group of patients and a group of primary and specialized care professionals.
* The control group will not receive any specific intervention. They receive usual care according to actually clinical practice guidelines.

Measurements:

* Main Variable: Patient Activation Measure questionnaire. This questionnaire values activation in patients with chronic diseases. It consists of 13 items that evaluate people's knowledge, skills and confidence in self-care for their health and medical care. Measured by a scale type Likert 1-4 with a total score between 0 and 100. 0 is the worst puntuation and 100 is the best puntuation.
* Knowledge about the disease, assessed through a self-administered self-made questionnaire. The questionnaire will measure the level of knowledge about secondary prevention of cardiovascular disease and will be based on the Questionnaire of Factors of Risk Cardiovascular previous translation-back translation and adaptation to the Spanish population.
* Attitude of the patient, measured from the self-administered self-efficacy Managing Chronic Disease Scale questionnaire . This questionnaire was developed to assess the self-efficacy or confidence perceived by the person to perform self-care activities for the management of their chronic disease. Includes 6 items with aspects such as fatigue, emotions and treatment with response from 1 (no confidence) to 10 (totally confident); the average final score of all the items is calculated (the higher the score, the more self-efficacy). This questionnaire has been translated into Spanish and used in our context in people with heart failure
* Adhesion to the Mediterranean diet from the Mediterranean Diet questionnaire It is a set of 14 short questions whose evaluation aims to provide information on adherence to the Mediterranean diet pattern. Scores below 7 indicate low adherence; Scores above 10 indicate good adherence. It has been validated in the Spanish population in the PREDIMED study .

International Physical Activity Questionnaire. This questionnaire has been used in several international studies and its validity has been evaluated recommending its use in different countries and languages The short version provides information on the time spent walking, in activities of moderate and vigorous intensity and in sedentary activities. Evaluates three specific characteristics of the activity: intensity (mild, moderate, vigorous), frequency (measured in days per week) and duration (time per day). After calculating the physical activity index, whose value corresponds to the product of the intensity (in METS) by the frequency, and by the duration of the activity) the patients are classified into three categories: low, medium and high.

Depression - Patient Health Questionnaire-9 .It is an instrument that not only allows detecting people with depressive disorder, but also allows to define the severity of the condition and to follow up on these people. It has been validated to Spanish demonstrating behavior similar to the original in English and a good acceptance by patients . It is a short instrument, designed to be self-administered. It consists of 9 items that assess the presence of depressive symptoms (corresponding to the DSM-IV criteria) present in the last 2 weeks. Each item has a severity index corresponding to: 0 = "never", 1 = "some days", 2 = "more than half of the days" and 3 = "almost every day".

Anxiety - Hospital Anxiety and Depression Scale. This scale is a 14-item questionnaire that was initially designed for the evaluation of anxiety and depression in non-psychiatric outpatient hospital services. It is a useful instrument validated in our setting and of special interest and usefulness in the context of PA. It is a measure composed of two sub-scales (Hospital Anxiety and Depression - A and Hospital Anxiety and Depression - D), of seven items each that are scored from 0 to 3. The authors recommend the points of 8 for possible cases and> 10 for cases probable in both sub-scales. One of its main virtues is the suppression of somatic symptoms so that it can be evaluated independently of the underlying somatic disease. However, in patients with coronary artery disease, it has been found that it underestimates people with depression , while the Hospital Anxiety and Depression - A sub-scale has a good specificity and predictive value to measure anxiety in this context.

Adherence to medication: Will be assessed with the Adherence Refill and Medication Adherence Scale (ARMS-e), validated in Spain and used to measure adherence to medication in patients with chronic diseases. It consists of 12 questions and there is no cut-off point, the lower the score, the better the adherence. To quantify adherence, a value of 1 to 4 (never, sometimes, almost always or always) is assigned to each of the responses according to a Likert-type scale.

Quality of life related to health - E5-5D-5L The EQ-5D, developed by the EuroQol Group (www.euroqol.org), is a generic and standardized instrument designed to describe and assess the quality of life related to health in both relatively healthy individuals (general population) and in groups of patients with different pathologies. It has been prepared in several languages, including Spanish, and used in various contexts, including the PA . The EQ-5D was born to try to offer a measure of self-perceived health that incorporated the individual preferences (utilities) on health status and that would serve as a measure of effectiveness in the economic evaluation of health technologies and health policies. It allows to reflect the quality of life associated with health, with the amount of life and offer a value of the gains in health, the Quality Adjusted Life Year (QALY). It consists of 2 parts: the person assesses their state of health, first in levels of severity by dimensions (descriptive system) and then in a visual analog scale (EVA) of more general evaluation. A third element of the EQ-5D is the index of social values obtained for each health state generated by the instrument. The descriptive EQ-5D system comprises 5 dimensions (mobility, personal care, daily activities, pain / discomfort and anxiety / depression). In the EVA the individual scores his health between two extremes, 0 and 100, worse and better state of health imaginable. The EQ-5D is available in two versions for adults, with 3 levels and 5 levels of response options, EQ-5D-3L and EQ-5D-5L, respectively. The EQ-5D-5L has shown to be a valid extension of the EQ-5D-3L that improves the measurement properties.

Use of health resources through a self-administered questionnaire contrasted with Clinical History information: visits to the doctor and / or nurse in the last 3 months, hospital admissions during the intervention, temporary or permanent ITs (number and time).

Explanatory and adjustment variables:

Of the patient (first level): Sociodemographic: age, sex, nationality, Autonomous Communities of residence, marital status (married / couple, single, separated, divorced, widowed), educational level (incomplete primary studies, complete primary education, education secondary school, university studies or equivalent), lives alone (yes / no), current occupation; Morbidity: type (stable angina, unstable angina, AMI), duration of ischemic heart disease (months), ventricular ejection fraction (≤ 35%,> 35%), classification of the New York Heart Association (I-IV), number and description of chronic concomitant diseases (O'Halloran list (63)); Treatment: pharmacological (acetylsalicylic acid or clopidogrel, beta-blockers, statins, other treatments), participation in a cardiac rehabilitation program before and during the study period (yes / no). This information will be collected from a self-administered self-prepared questionnaire contrasted with information from the Clinical History.

Clinics: blood pressure, body mass index (BMI), lipid profile (HDL-C, LDL-C), smoking habit, number and frequency of anginal episodes. These variables will be collected through a self-administered self-prepared questionnaire contrasted with information from the Clinical History.

Analysis

An analysis of multilevel mixed models is proposed for the main result, where the response variable will be the difference between the final and initial score obtained in the attitude questionnaire administered to the participating professionals and the explanatory variable will be the dichotomous intervention variable (1 = Virtual Community of Practice / 0 = Control). This model will consider the co-variables age, sex and clinical characteristics of the patient with Heart Disease and will take into account the random effect associated with Primary Care Centre. To control a possible selection bias and increase the accuracy of the model, the Propensity Score will be used. The analyzes will be carried out by intention to deal with the statistical software R Core Team (2014) http://www.R-project.org/ and Statistical Package for the Social Sciences 18.

Analysis: a linear regression model of mixed effects will be estimated to estimate the effect of participating in theVirtual Community of Practice. In addition, subgroup analyses will be carried out and indicators of the functioning of the Virtual Community of Practice will be measured through techniques of Social Network Analysis and Control Charts. There will be an economic evaluation of the Virtual Community of Practice from the perspective of the National Health System and from the social perspective.

ELIGIBILITY:
Inclusion Criteria:

* Active diagnosis of ischemic heart disease in the year prior to inclusion in the study; have Internet at home or phone
* be able to follow the requirements of the study
* having signed informed consent for participation in the study.

Exclusion Criteria:

* low probability of cooperation in the study
* bystanders or displaced status
* institutionalized, with a terminal illness, physical or mental disability that prevents respond to questionnaires properly.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

PRIMARY OUTCOMES:
Patient Activation Measure questionnaire | Patient Activation Measure measured at 18 months
  It has 13 items, measured with a Likert scale (from 1 to 4). This questionnaire values activation in patients with chronic diseases. It evaluates people's knowledge and skills in self-care. Puntuation is 0 to 100 (best puntuation)

CONTACTS AND LOCATIONS:
Locations (1):
- Sofía Garrido elustondo, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be collected from self-reported questionnaires and the electronic medical records.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 18 months
Access Criteria: Only researchers can Access to the study data.

REFERENCES:
- [Background] Hibbard JH, Greene J. What the evidence shows about patient activation: better health outcomes and care experiences; fewer data on costs. Health Aff (Millwood). 2013 Feb;32(2):207-14. doi: 10.1377/hlthaff.2012.1061. PMID 23381511
- [Background] Mosen DM, Schmittdiel J, Hibbard J, Sobel D, Remmers C, Bellows J. Is patient activation associated with outcomes of care for adults with chronic conditions? J Ambul Care Manage. 2007 Jan-Mar;30(1):21-9. doi: 10.1097/00004479-200701000-00005. PMID 17170635
- [Background] Salvado-Hernandez C, Cosculluela-Torres P, Blanes-Monllor C, Parellada-Esquius N, Mendez-Galeano C, Maroto-Villanova N, Garcia-Cerdan RM, Nunez-Manrique MP, Barrio-Ruiz C, Salvador-Gonzalez B; en representacion del grupo de investigacion del proyecto COIB 5367-11. [Heart failure in primary care: Attitudes, knowledge and self-care]. Aten Primaria. 2018 Apr;50(4):213-221. doi: 10.1016/j.aprim.2017.03.008. Epub 2017 Jun 23. Spanish. PMID 28652033
- [Derived] Vall-Roque H, Ramos-Garcia V, Rivero-Santana A, Torres-Castano A, Cifuentes P, Koatz D, Garcia-Garcia J, Pacheco-Huergo V, Rello P, Santos-Alvarez A, Campillejo Garcia A, Garrido Elustondo S, Sanmartin M, Perestelo-Perez L, Gonzalez-Gonzalez AI, Orrego C. A virtual community of practice to empower patients with recent ischemic heart disease: A randomized controlled trial. Health Psychol. 2025 Jun;44(6):630-642. doi: 10.1037/hea0001439. Epub 2024 Dec 16. PMID 39679979
- [Derived] Gonzalez-Gonzalez AI, Perestelo-Perez L, Koatz D, Ballester M, Pacheco-Huergo V, Ramos-Garcia V, Torres-Castano A, Rivero-Santana A, Toledo-Chavarri A, Valcarcel-Nazco C, Mateos-Rodilla J, Obaya-Rebollar JC, Garcia-Garcia J, Diaz-Sanchez S, Morales-Cobos L, Bosch-Fontcuberta JM, Vallejo-Camazon N, Rodriguez-Almodovar A, Del Castillo JC, Munoz-Balsa M, Del Rey-Granado Y, Garrido-Elustondo S, Tello-Bernabe ME, Ramirez-Puerta AB, Orrego C. Effectiveness and cost-effectiveness of a virtual community of practice to improve the empowerment of patients with ischaemic heart disease: study protocol of a randomised controlled trial. BMJ Open. 2020 Oct 12;10(10):e037374. doi: 10.1136/bmjopen-2020-037374. PMID 33046465